CLINICAL TRIAL: NCT05300074
Title: Equivalence Test of Two Different Inspiratory Muscle Training Protocols: a Randomised Controlled Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: adjustments needed after pilot period and delay because of reduced staff
Sponsor: Spinal Cord Injury Centre of Western Denmark (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-378-21
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-11

CONDITIONS: Inspiratory Muscle Training
Keywords: IMT; Maximal inspiratory pressure; MIP

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training two times per week (Experimental): Training two times per week. IMT with 5 rounds and 12 repetitions in each round at 60-80% MIP. The primary protocol will end at 6 weeks and the self-administered long-term protocol will end at 12 months after intervention start.
  Interventions: Other: Inspiratory Muscle Training
- Training five times per week (Experimental): Training five times per week. IMT with 5 rounds and 12 repetitions in each round at 60-80% MIP. The primary protocol will end at 6 weeks and the self-administered long-term protocol will end at 12 months after intervention start.
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — IMT is performed with an IMT Threshold flute that can be adjusted according to the MIP. The training resistance start at 60% MIP and is calculated weekly and end (if tolerated) at 80 % MIP.

SUMMARY:
The objective of this study is to investigate if six weeks of high intensity Inspiratory Muscle Training (IMT) performed two times a week has the same effect as five times a week in hospitalized patients with first time Spinal Cord Injury (SCI).

Design/ methods: A Randomised controlled trial (RCT) including 60 patients, with reduced Maximal Inspiration Pressure (MIP) will be recruited at two specialized SCI centers in Denmark. Primary outcome is MIP after six weeks of training. Secondary outcome will be reported on Rating Perceived Exertion (RPE), voice performance, Quality Of Life (QOL)and sleep quality. Furthermore, long term follow-up at 12 months after start of intervention will also be performed.

DETAILED DESCRIPTION:
Background: SCI may result in various disabilities including both physical, cognitive, emotional and social domains. Motor function and function of the respiratory muscles are often decreased and may influence the patient's activities of daily activities and QOL. IMT is training to improve the strength and endurance of diaphragm and the external intercostal muscles. Various training protocols of IMT have shown efficient to increase lung function. Although, a recent meta-analysis suggest that high intensity training may be more efficient it is less clear at what weekly frequency IMT should be performed.

Thus, the objective of this study is to investigate if six weeks of high intensity IMT performed two times a week has the same effect as five times a week in hospitalized patients with first time SCI.

Design/ methods: A Randomised controlled trial (RCT) including 60 patients, with reduced MIP will be recruited at two specialized SCI centers in Denmark. Primary outcome is MIP after six weeks of training. Secondary outcome will be reported on end of treatment and long term follow-up (12 months after start of intervention) in RPE, voice performance, QOL and sleep quality. The two intervention arms will consist of one arm training two times a week and the other arm training five times a week. The training protocol in both arms will include five rounds of IMT with 12 repetitions at 60 % of MIP. MIP will be increased 10 % every week if tolerated by the patient until 80 % of MIP is reached. After six weeks patients are motivated to continue training by themself up to 12 months after start of intervention.

ELIGIBILITY:
Inclusion Criteria:

* First time SCI within 0-6 months
* Age ≥ 18 years
* Neurological level: C4 -TH12 and C1-C4 (AIS D only)
* Severity/ AIS: A, B, C or D
* Able to give informed concent and understand and read Danish
* Mental able to understand and participate in a lung function assessment
* Decreased MIP according to normal gender and age adjusted MIP values

Exclusion Criteria:

* Lung disease or lung infection at the time of inclusion
* Co-morbidity or other contra indications
* Injury that hinder mouth shutting
* Respirator or tracheal tube use
* Experience of severe dizziness or vomiting during training
* Not expected to be hospitalised for at least 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | Change from baseline assessment (0-4 days before treatment start) to End of treatment assessment (6 weeks after intervention start)
  MIP is an objective measurement that indirectly describe the inspiratory muscle strength

SECONDARY OUTCOMES:
Rating of Perceived Exertion | Baseline assessment (0-4 days before treatment start), End of treatment assessment (6 weeks after intervention start) Longterm follow up (12 months after intervention start)
  RPE is a way of measuring physical activity intensity level. RPE will be reported in regard to the IMT training and will express the experience of how hard the IMT was feelt.
Voice performance | Baseline assessment (0-4 days before treatment start), End of treatment assessment (6 weeks after intervention start) Longterm follow up (12 months after intervention start)
  The voice performance is measured with voice volume recording of an a-sound with the App Voice Analyst along with phonation endurance.
Experienced quality of life measured with the The basic Spinal cord injury (SCI) Data Set for Qualify of Life | Baseline assessment (0-4 days before treatment start), End of treatment assessment (6 weeks after intervention start) Longterm follow up (12 months after intervention start)
  The basic SCI Data Set for Qualify of Life consists of QOL measured by three domains; overall, physical and mental QOL. Each domain is subjectively rated on a 0-10 scale, with 0 = completely dissatisfied and 10 = completely satisfied.
Experienced sleep Quality measured with Pittsburgh Sleep Quality Index (PSQI) tool | Baseline assessment (0-4 days before treatment start), End of treatment assessment (6 weeks after intervention start) Longterm follow up (12 months after intervention start)
  Sleep quality is measured by sleep quality experience and report of circumstances that may influence sleep. The global PSQI score is calculated by totaling the seven component scores (Each weighted on a 0-3 interval scale), providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Maximal inspiratory pressure | Change from baseline assessment (0-4 days before treatment start) to longterm follow up (12 months after intervention start)
  MIP is an objective measurement that indirectly describe the inspiratory muscle strength
Patients' Global Impression of Change (PGIC) scale | collected at 6 week and 12 months after start of the intervention
  Patient reported outcome at follow up. Scores from 0 to 6, with 0 reporting no change and 6 aa significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Erhard T. Næss-Schmidt, PhD, Principal Investigator — Spinal Cord Injury Centre of Western Denmark
Locations (1):
- Spinal cord injury center Western Denmark, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No
no plan